CLINICAL TRIAL: NCT00740688
Title: The Effects of Logan Basic Technique on Bilateral Weight Balance
Brief Title: Basic and Balance: Logan Basic Technique on Bilateral Weight Balance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Logan College of Chiropractic (Other)
Responsible Party: Patrick Montgomery, DC, Logan University, College of Chiropractic
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: SR0225080130
Record Dates: First submitted 2008-08-21; First posted 2008-08-25 (Estimated); Last update posted 2008-08-25 (Estimated); Status verified 2008-08

CONDITIONS: Pelvic Adjusting (LBT)

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (Experimental): A Logan Basic Apex Contact, which is a contact that is placed on the anterior surface of the sacrotuberous ligament with a light force directed posterior with varying degrees of laterality.
  Interventions: Procedure: Logan Basic Apex Contact
- Sham Group (Sham Comparator): light force contact applied to the inferior surface of the sacrotuberous ligament, directed straight superiorly.
  Interventions: Procedure: Sham Logan Basic apex contact

INTERVENTIONS:
Procedure: Logan Basic Apex Contact — A Logan Basic Apex Contact, which is a contact that is placed on the anterior surface of the sacrotuberous ligament with a light force directed posterior with varying degrees of laterality.
  Arms: Experimental Group
Procedure: Sham Logan Basic apex contact — light force contact applied to the inferior surface of the sacrotuberous ligament, directed straight superiorly.
  Arms: Sham Group

SUMMARY:
This is an experimental study to examine whether a chiropractic intervention (specifically Logan Basic Technique) can help restore balance distribution in individuals with or without vertebral subluxations.

DETAILED DESCRIPTION:
Postural imbalance caused by abnormal weight distribution in the body may cause discomfort, pain and deformity. In the human body, weight and the resistance to gravity is controlled by the bones that make up the skeletal system which are supported by ligaments and tendons. Without this framework holding up upright, we would fall to the ground due to the external forces of gravity. When one half of the body must work harder to support more weight than the other, the half of the body with the greater imbalance may become strained. As a result of the imbalance, strain and tension will increase causing a decrease in blood supply which will decrease proper exchange of wastes, nutrients, and oxygen causing an increase in toxicity. According to the Logan Basic Methods textbook, as long as there remains a symptom of strain in muscle tissue as a result of abnormalities of the body framework, such a muscle is capable, with slight assistance, of restoring its subluxated attachments to their normal relationship. The slightest force exerted on either of its attachments, directly or indirectly, tends to approximate its points of attachment and result in a decreased strain of the muscle. Therefore, the necessary amount of force applied to improve postural distortion is dependent upon the nature or degree of the patient's postural distortion or muscular imbalance.

The system of Logan Basic Methods uses structural analysis from radiography combined with postural and clinical examination findings to determine and apply specific low-force adjustments to the pelvis and spine. The most commonly applied contact of Logan Basic Technique, the apex contact, specifically contacts the sacrotuberous ligament, which connects the ischial tuberosity to the anterior aspect of the sacrum, as it attaches to the sacrum. This ligament is believed to play an integral role in the stability of the pelvis, especially during nutation and counter-nutation. This is further evidenced by a study of the function of the long dorsal sacroiliac ligament, of which the sacrotuberous ligament played a significant role in counter-balancing the pelvis during nutation and counter-nutation.

The Midot Postural Analyzer QPS-200 provides data regarding weight distortion of the actual body weight within a 360 degree radius, in a two dimensional plane.

Similar studies have been performed by Logan students in the past. The first study found, from 1990, was designed as a double blind study with apex contacts or sham adjustments given to participants in an attempt to determine affects of Logan Basic Technique on leg length deficiency and balance. Only one adjustment was given to each participant. Results were inconclusive, with no favorable results for the intervention. Another similar study performed in 1996 by Goutlet, Webb, and Lawson under the guidance of Dr. Brian Snyder was a double blind study that used an apex contact for the experimental intervention and a sham adjustment for the control group. The researchers used two common bathroom scales for their data collection. A positive correlation was found between the weight distribution changes pre-post adjustment in the experimental group, with only one treatment given to subjects in the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be limited to Logan College of Chiropractic students.
* Have an initial imbalance in their weight distribution of greater than 4 pounds.

Exclusion Criteria:

* Pregnant
* Persons with an imbalanced structural scoliosis, which will be determined by the utilization of a posterior plumb line.
* Taking herbs or medication that affects balance
* Individuals with problems maintaining their balance as seen in Meniere's syndrome, otitis interna and otitis media
* Individual diagnosed Diabetes
* Individuals currently receiving any spinal manipulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2008-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
weight distribution | before and after treatment, 3 times over 3 days

SECONDARY OUTCOMES:
center of gravity | before and after treatment, 3 times over 3 days